CLINICAL TRIAL: NCT06147284
Title: MOVIN' CARE for PD: A Project on Community Awareness, Rehabilitation and Empowerment for Parkinson's Disease (Risk Management)
Brief Title: MOVIN' CARE for PD (Risk Management)
Acronym: jcpdmcP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Society for Rehabilitation (Other); The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EA230262P
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-09

CONDITIONS: Parkinson's Disease (At-risk Cases)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Due to the nature of this trial, neither the staff, participants nor care provider can be masked to allocation. The data analyst will be blinded after study completion by having the intervention group information coded. All outcome assessors will be blinded to subject allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional exercise (Experimental): This is an intervention with six 90-minute sessions. Progressive traditional exercise including warm-up exercises, resistance training, stretching routines, and cool-down exercises will be introduced. Both face-to-face and home-based online modes of delivery are available.
  Interventions: Behavioral: Preventive interventions
- Yoga intervention (Experimental): The intervention, comprising six 90-minute sessions, will be delivered by a trained mindful yoga instructor in group format. The intervention is based on our previously tested mindfulness yoga programme for people with PD (31). Following a universal Hatha Yoga practice, the session comprises mindfulness practice of yoga sequence, breathing exercise, and guided meditation. Both face-to-face and home-based online modes of delivery are available.
  Interventions: Behavioral: Preventive interventions
- Arts-based intervention (Experimental): Participants in the six 90-minute sessions in this intervention will be engaged in art-making processes through multiple art modalities such as visual arts, dance/ movement, music, drama, and creative writing. Each section is usually structured with Filling-in - greetings and check-in, Bridging - warm-up, Decentering - arts making and appreciation, Harvesting - sharing and response, and Closure. Both face- to-face and home-based online modes of delivery are available.
  Interventions: Behavioral: Preventive interventions
- Somatic intervention (Experimental): The intervention involves six 90-minute sessions led by a trained somatic practitioner in group format. Participants will be guided to bring awareness to their body and to connect with their internal sensations through exploring imageries related to their somatic experiences. They will also learn some somatic techniques that enable them to use their bodies more effectively. Both face-to-face and home- based online modes of delivery are available.
  Interventions: Behavioral: Preventive interventions

INTERVENTIONS:
Behavioral: Preventive interventions — Parallel randomized controlled trial

SUMMARY:
The goal of this intervention study is to investigate the effectiveness of three preventive interventions - yoga, arts-based approaches, and somatic practices, with reference to an active control group - traditional exercises, in enhancing psycho-social-spiritual well-being among people at risk of Parkinson's disease (Parkivers). The hypotheses include:

H1: Yoga, arts-based, somatic interventions will significantly improve the psycho-social- spiritual wellbeing (i.e., perceived stress, anxiety and depressive symptoms, and quality of life) among Parkivers H2: In comparison to traditional exercise, yoga, arts-based, and somatic interventions will have a significant effect on psycho-social-spiritual well-being among Parkivers H3: Yoga, arts-based, somatic, and traditional exercise training interventions will have a significant effect in reducing PD-related motor symptoms H4: Yoga, arts-based, somatic interventions have a significant long-term effect on improving psycho-social-spiritual well-being among Parkivers

Eligible participants will be invited to undergo baseline assessments before randomization to attend a six-session intervention group. To investigate the immediate and long-term effect of the preventive measures, repeated outcome measures will be conducted at six time-points: A baseline assessment prior to randomization (T0), and follow-ups at 2-months (T1), 6-months (T2), 12-months (T3), 18- months (T4), 24-months (T5).

DETAILED DESCRIPTION:
Parkinson's disease (PD), the second most common neurodegenerative disease, usually results in physical deterioration, as well as a spectrum of psychosocial sequels that could bring various challenges on one's daily lives. Patients experience common motor symptoms, including tremor, rigidity, bradykinesia, and postural instability, in parallel with psychosocial stressors (i.e., non- motor symptoms NMS), such as sleep disturbance, cognitive deficits, gastrointestinal symptoms, dopaminergic drug-induced behaviors (e.g., hallucination, impulse control issues) and mood disturbance (e.g., depression, anxiety). While 21% of individuals struggling with the disease reported at least one of these psychosocial symptoms within the initial stage of the disease, they are generally at risk for increased emotional distress, cognitive declines, and elevated stress hormone (cortisol) levels.

Both motor and non-motor symptoms of Parkinson's disease could affect the quality of life of individuals and that of their caregivers. A cross-sectional study conducted by our research team has explored the symptom burden and support care needs in people with PD across East and Southern Asia (n=186), revealing significant unmet needs among Hong Kong PD patients regarding their psychosocial-spiritual concerns. In particular, they experience significant, moderate palliative care needs at the early to middle course of the illness. The extent of unmet support care needs among patients with mild to moderate PD is as great as that among patients with other chronic health conditions, such as advanced cancer, late-stage lung cancer, stage 4/5 chronic obstructive pulmonary disease and late stage chronic kidney disease. The visible and unpredictable symptoms of a distorted body (e.g., tremor and gait dysfunction) and the suppressed expressions due to having a masked face, reduced voice and slurred speech often results in difficulty seeking help and stigmatization of the disease.

Despite the tremendous influences and common occurrence of NMS, they are surprisingly under- recognized in clinical practice because of the lack of spontaneous verbal complaints by the patients, as well as the lack of systematic questioning by healthcare professionals. A qualitative exploration of the illness experience of local PD patients highlighted the importance and urgent need for holistic PD interventions that emphasizes on early identification and preventive measures of individual who are at risk for PD patients, alleviation of the effects of the psychological sequels to PD patients, as well as the reduction of stigma and promotion of community support towards PD.

The study adopts a 4-arm randomized controlled design, aiming to investigate the effectiveness of three preventive interventions - yoga, arts-based approaches, and somatic practices, with reference to an active control group - traditional exercises, in enhancing psycho-social-spiritual well-being among people at risk of PD.

ELIGIBILITY:
Inclusion Criteria:

* adults who are aged 18 or above
* able to give written informed consent
* able to have access to the Internet and a smartphone/tablet/laptop
* willing to download mobile apps related to the research project
* able to comprehend Chinese.

Exclusion Criteria:

* significantly cognitive impaired (indicated by Abbreviated Mental Test lower than 6)
* engaged in regular instructor-led mind-body exercise (e.g., Taichi), expressive arts therapy, or somatic practices (>2 times per week) in the past 3 months)
* currently participating in any other behavioral or pharmacological trial
* with other contradiction(s) that may limit their full participation (e.g. severe hearing or vision impairment, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-11 (Estimated)

PRIMARY OUTCOMES:
Change of Perceived stress level | A baseline assessment prior to randomization (T0), and follow-ups at 2-months (T1), 6-months (T2), 12-months (T3), 18- months (T4), 24-months (T5).
  Perceived Stress Scale (PSS) uses a five-point Likert scale to measure the perceived stress level. The 10 items in the scale can be divided into two subscales, measuring the perceived helplessness, and inadequacy of self-efficacy. A high score indicates a high perceived stress level. The Cronbach's α of the validated Chinese version of the scale is 0.85.
Change of Quality of Life | A baseline assessment prior to randomization (T0), and follow-ups at 2-months (T1), 6-months (T2), 12-months (T3), 18- months (T4), 24-months (T5).
  The brief World Health Organization Quality-of-Life Scale (WHOQOL-BREF) will measure the four dimensions of quality of life, including physical health, psychological health, social relationships, and environment. The scale consists of 26 items and uses a five-point Likert scale. The higher the score, the better the quality of life. The Cronbach's α of the subscales ranges from 0.73-0.82.

SECONDARY OUTCOMES:
Change of PD-related motor and non-motor symptoms | A baseline assessment prior to randomization (T0), and follow-ups at 2-months (T1), 6-months (T2), 12-months (T3), 18- months (T4), 24-months (T5).
  PD-related motor and non-motor symptoms will be measured by the validated Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS- UPDRS)(Chinese) Part I to IV [13]. The four dimensions measured by the scale include (i) non-motor experiences of daily living, (ii) motor experiences of daily living, (iii) severity of motor symptoms, and (iv) motor complications. High scores indicate great disease severity. Cronbach's α are 0.79-0.94. In addition, Mon4t (by Montfort Brain
  Monitor, Tel-Aviv, Israel) is a mobile application that evaluates PD-related motor symptoms of participants. It is commonly used for tasks including timed-up-and-go, finger tapping, measuring resting tremor and postural tremor.
Change of Anxiety and depressive symptoms | A baseline assessment prior to randomization (T0), and follow-ups at 2-months (T1), 6-months (T2), 12-months (T3), 18- months (T4), 24-months (T5).
  Anxiety and depressive symptoms will be measured by the Hospital Anxiety and Depression Scale (HADS). The 14 scale items are evenly divided into anxiety (7 items) and depression (7 items). The scale uses a four-point Likert scale. A high score indicates severe psychological distress. Cronbach's α is 0.86.
Change of Constipation severity | A baseline assessment prior to randomization (T0), and follow-ups at 2-months (T1), 6-months (T2), 12-months (T3), 18- months (T4), 24-months (T5).
  Constipation severity will be measured by the 16-item Chinese version of the Constipation severity instrument (CSI) (Cronbach's α is 0.93-0.95). It consists of three subscales, namely the obstructive defecation, colonic inertia, and pain. The higher the score, the higher the constipation severity (total scores 0-78).
Change of Bowel habits | A baseline assessment prior to randomization (T0), and follow-ups at 2-months (T1), 6-months (T2), 12-months (T3), 18- months (T4), 24-months (T5).
  Bowel habits will be measured by a self-reported 7-day bowel diary to document the number of bowel movements, sensation of complete bowel emptying, stool consistency rated on the Bristol Stool Form Scale, and the use of laxatives (type and frequency).
Change of Gut microbiota composition | A baseline assessment prior to randomization (T0), and follow-ups at 2-months (T1), 6-months (T2), 12-months (T3), 18- months (T4), 24-months (T5).
  Fresh stool samples will be collected to investigate participants' gut microbiota composition. Shotgun metagenomics sequencing of the fecal samples will be conducted using the DNBseqTM sequencing platform with a 100 bp paired-end protocol by BGI Tech Solutions (Hong Kong) Co., Ltd. The microbiota composition will be documented by the MetaPhlan3.
User's satisfaction | 2-months (T1)
  User's satisfaction of the intervention will be measured by 11 items on a five- points Likert scale. The scale will be used to understand the participant's satisfaction and perceived effectiveness of the preventive intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rainbow T.H. Ho, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- 2/F., The Hong Kong Jockey Club Building for Interdisciplinary Research, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No